CLINICAL TRIAL: NCT05332457
Title: The Effect of Beta-blocker on Chronotropic Response and Cardiorespiratory Fitness in Patients With Atrial Fibrillation: a Crossover Randomized Controlled Trial.
Brief Title: The Effect of Beta-blocker on Chronotropic Response and Cardiorespiratory Fitness in Patients With Atrial Fibrillation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202201028MINB
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Beta-blocker; Chronotropic response; Cardiorespiratory fitness
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-centered, crossover, randomized (1:1) study.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor are blinked to participants' allocation group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Phase I : Participants will undergo first CPET (Day 0) at trough concentration of BB. After 7-day regular usage of BB, the second CPET(Day 7) will be performed at peak concentration of BB. Participants will enter the second phase if the results of CPET fulfill the pre-determined conditions as follows: (1) Chronotropic index < 0.8 at peak level of BB, (2) Resting HR < 110 bpm at trough level of BB, (3) Absent of unstable arrhythmia or unstable hemodynamics during CPET at trough level.
  Phase II: BB dosage will be reduced. Daily blood pressure, heart rate and adverse event will be recorded. If participants remained clinically stable, the third CPET(Day 21) will be performed 14 days after the reduction of dosage. If participants' resting heart rate exceed 110 bpm, the dosage will be adjusted to the original level.
  Interventions: Drug: Reduced dosage of beta-blocker
- Arm B (Active Comparator): Phase I : Participants will undergo first CPET(Day 0) at peak concentration of BB. After 7-day regular usage of BB, the second CPET(Day 7) will be performed at trough concentration of BB. Participants will enter the second phase if the results of CPET fulfill the pre-determined conditions as follows: (1) Chronotropic index < 0.8 at peak level of BB, (2) Resting HR < 110 bpm at trough level of BB, (3) Absent of unstable arrhythmia or unstable hemodynamics during CPET at trough level.
  Phase II: BB dosage will be reduced. Daily blood pressure, heart rate and adverse event will be recorded. If participants remained clinically stable, the third CPET(Day 21) will be performed 14 days after the reduction of dosage. If participants' resting heart rate exceed 110 bpm, the dosage will be adjusted to the original level.
  Interventions: Drug: Reduced dosage of beta-blocker

INTERVENTIONS:
Drug: Reduced dosage of beta-blocker — Phase I:
  1. CPET performed at trough BB concentration: participants will undergo CPET at least 30 hours after last beta-blocker usage.
  2. CPET performed at peak BB concentration : participants will undergo CPET at 3 hours after last beta-blocker usage.
  Phase II:
  BB dosage will be reduced.

SUMMARY:
This is a prospective study to evaluate changes in exercise capacity and chronotropic response to exercise before and after beta-blocker dosage reduction in patients with atrial fibrillation (AF).

DETAILED DESCRIPTION:
Rate control therapy is the first-line treatment for atrial fibrillation (AF). Resting heart rate(HR) is the treatment target of rate control therapy in current clinical practice; However, the optimal value for resting heart rate in AF remained unclear. Beta-blocker(BB) is widely used as rate-control agent. It is concerned that excessive use of BB might lead to a negative effect on exercise capacity in patients with AF. The aim of this study is to explore the effect of Beta-blocker on hemodynamic parameters and peak oxygen uptake during cardiopulmonary exercise test (CPET).

ELIGIBILITY:
Inclusion Criteria:

1. > 20 years of age.
2. Clinically stable patients with persistent atrial fibrillation using beta-blocker as rate-control agent without dosage adjustment for at least 3 months.
3. Resting heart rate < 80 bpm.
4. Left ventricular ejection fraction > 50%.

Exclusion Criteria:

1. Beta-blocker usage due to indications other than rate control for atrial fibrillation.
2. Inability to perform a cardiopulmonary exercise testing.
3. Presence of contraindications for cardiopulmonary exercise testing according to the American College of Sports Medicine's Guidelines for Exercise Testing and Prescription.
4. Patients with implantable cardioverter defibrillator or pacemaker.
5. Pregnancy.
6. Inability to provide informed consent.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen intake | The change in peak oxygen uptake will be measured at day 0 , day 7 and day 21.
  Peak oxygen intake will be assessed with symptom-limited cardiopulmonary exercise testing.
Chronotropic response to exercise | The change in chronotropic response to exercise will be measured at day 0 , day 7 and day 21.
  Plasma norepinephrine level was obtained before and immediately after cardiopulmonary exercise testing to assess the relationship of beta-blocker, circulating norepinephrine level and chronotropic response to exercise.

SECONDARY OUTCOMES:
European Heart Rhythm Association (EHRA) symptom scale | The change in European Heart Rhythm Association (EHRA) score will be measured at day 0 , day 7 and day 21.
  The investigators will assess the change in EHRA symptom scale. The EHRA score ranges from 1 to 4. Higher scores indicate more severe symptoms.
Cardiac output and stroke volume | The change in cardiac output and stroke volume will be measured at day 0 , day 7 and day 21.
  Cardiac output and stroke volume during incremental exercise testing will be assessed by impedance cardiography.
Cognitive function | The change in MoCA will be measured at day 0 , day 7 and day 21.
  The investigators will assess the change in Montreal Cognitive Assessment (MoCA). The total score of MoCA ranges from 0 to 30. Higher scores indicate better cognitive function.
NT-proBNP | The change in NT-proBNP will be measured at day 0 , day 7 and day 21.
  NT-proBNP level will be assessed before and immediate after the cardiopulmonary exercise test.
Quality of life evaluation | The change in SF-36 will be measured at day 0 , day 7 and day 21.
  The investigators will assess the change in 36-Item Short Form Survey (SF-36). SF-36 consists of eight domains of health status. The score of each domain ranges from 0 to 100. Higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Jui Chuang, MD, Principal Investigator — Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No